CLINICAL TRIAL: NCT01660152
Title: Analysis of Technique Comparison With a Vacuum Erection Device as Part of an Erectile Rehabilitation Program Following Robotic Radical Prostatectomy: A Randomized Comparison of Methodology
Brief Title: Vacuum Erection Device in Improving Recovery of Erectile Function in Patients With Prostate Cancer Undergoing Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-11019; NCI-2012-00997 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Male Erectile Disorder; Prostate Cancer; Sexual Dysfunction
Keywords: male erectile disorder; prostate cancer; Laparoscopic prostatectomy
MeSH Terms: conditions — Erectile Dysfunction; Prostatic Neoplasms; Sexual Dysfunction, Physiological | interventions — Menogaril; methyl 3-mercaptopropionimidate; Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (vacuum therapy, holding erection for 2 minutes) (Experimental): Patients receive daily vacuum therapy over 10 minutes while holding erection for 2 minutes after undergoing RALP. Patients complete erection process 5 times. SHIM questionnaire administration will be completed prior to surgery and at 3, 6, 12 months and the compliance questionnaire at 3, 6, 12 months.
  Interventions: Other: Sexual Health Inventory for Men (SHIM) questionnaire administration; Procedure: management of therapy complications; Procedure: Daily vacuum therapy
- Group B (vacuum therapy, holding erection for 5 minutes) (Experimental): Patients receive daily vacuum therapy over 10 minutes while holding erection for 5 minutes after undergoing RALP. Patients complete erection process 2 times.Patients complete erection process 5 times. SHIM questionnaire administration will be completed prior to surgery and at 3, 6, 12 months and the compliance questionnaire at 3, 6, 12 months.
  Interventions: Other: Sexual Health Inventory for Men (SHIM) questionnaire administration; Procedure: management of therapy complications; Procedure: Daily vacuum therapy

INTERVENTIONS:
Other: Sexual Health Inventory for Men (SHIM) questionnaire administration — Questionnaire will be completed prior to surgery and at 3, 6, 12 months and the compliance questionnaire at 3, 6, 12 months.
  Other Names: assessment
Procedure: management of therapy complications — Receive VED
  Other Names: complications of therapy, management of
Procedure: Daily vacuum therapy — Patients randomized to Group A or Group B following removal of catheter at first post op visit following surger. Daily vacuum therapy for approximately 10 minutes. Depending on which group randomized to erection held for 2 minutes or 5 mintues.

SUMMARY:
The purpose of this study is to determine which technique in using a vacuum erection device (VED) is best. Erectile dysfunction (ED) after robotic prostate cancer surgery is a concern for both the surgeon and the patient. Recent studies have shown that beginning to use the vacuum pump on a daily basis starting with in 2-8 weeks may help prevent the start of penile shrinkage. This is a potential issue that can occur because of decreased blood flow after prostate cancer surgery. This study will allow researchers to determine and compare vacuum therapy techniques and erectile function outcomes of patients who have prostate cancer surgery

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine sexual function and penile morphometric outcomes for the post-robotic-assisted laparoscopic prostatectomy (RALP) patients undergoing daily vacuum therapy using one of two randomized methods and whether these outcomes differ.

SECONDARY OBJECTIVES:

I. Compare compliance rates between the two randomized groups using the compliance questionnaire and a diary collected from patients at each follow up visit.

II. Compare overall patient satisfaction with the recovery procedure between the two randomized groups utilizing the SHIM (Sexual Health Inventory for Men) questionnaire.

OUTLINE: Patients are randomized to 1 of 2 treatment groups.

GROUP A: Patients receive vacuum therapy daily over 10 minutes while holding erection for 2 minutes after undergoing RALP. Patients complete erection process 5 times.

GROUP B: Patients receive vacuum therapy daily over 10 minutes while holding erection for 5 minutes after undergoing RALP. Patients complete erection process 2 times.

After completion of study treatment, patients are followed up at 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active men without the consistent use of erectile aids pre-operatively (i.e. oral pharmacotherapy, intraurethral prostoglandin E1 [PGE1], intracavernosal injection therapy and penile implants)
* Undergoing a bilateral nerve sparing robotic prostatectomy
* Pre-operative baseline SHIM total score of greater than or equal to 17
* Presence of a female sexual partner
* Dexterity necessary to operate vacuum pump

Exclusion Criteria:

* Has a history of cardiac failure, angina, or life-threatening arrhythmia within the past 6 months
* Has taken or has been prescribed nitrate medication in any form in the last 6 months
* Has a known sensitivity to Phosphodiesterase type 5 inhibitors such as Sildenafil, Tadalafil or Vardenafil
* Men with sickle cell anemia
* Men with insufficient manual dexterity to operate vacuum device
* Men with a history of known penile deformity or Peyronie's disease
* Pre or postoperative androgen therapy
* Pre or postoperative radiation therapy to pelvic area
* Men actively smoking at time of enrollment, 1 pack per day or more

Max Age: 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-09; Primary Completion 2013-07-17 (Actual); Study Completion 2013-07-17 (Actual)

PRIMARY OUTCOMES:
Changes in sexual function based on the self reported SHIM assessment and penile morphometric outcomes based on penile dimension measurements at rest | 3 months post-surgery
  Summarized according to assigned treatment group. Linear mixed models will be used to model the changes over time.
Changes in sexual function based on the self reported SHIM assessment and penile morphometric outcomes based on penile dimension measurements at rest | 6 months post-surgery
  Summarized according to assigned treatment group. Linear mixed models will be used to model the changes over time.
Changes in sexual function based on the self reported SHIM assessment and penile morphometric outcomes based on penile dimension measurements at rest | 12 months post-surgery
  Summarized according to assigned treatment group. Linear mixed models will be used to model the changes over time.

SECONDARY OUTCOMES:
Compliance and overall patient satisfaction (1 to 25 point scale) based on the self reported compliance diary and SHIM questionnaires | Up to 12 months post-surgery
  Summarized according to assigned treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Ronney Abaza, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu